CLINICAL TRIAL: NCT03887780
Title: A Real-World, Prospective, Observational Study to Evaluate the Safety and Effectiveness of Rivaroxaban (Xarelto®) for Prevention of Stroke and Systemic Embolism in Indian Patients With Non-valvular Atrial Fibrillation (NVAF)
Brief Title: A Study to Evaluate the Safety and Effectiveness of Rivaroxaban (Xarelto) for Prevention of Stroke and Systemic Embolism in Indian Patients With Non-valvular Atrial Fibrillation (NVAF)
Acronym: XARIN
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Collaborators: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 20387
Record Dates: First submitted 2019-03-21; First posted 2019-03-25 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: Non-valvular Atrial Fibrillation (NVAF)
Keywords: Stroke;; Systemic embolism
MeSH Terms: conditions — Stroke | interventions — Rivaroxaban

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Treatment: Rivaroxaban treatment-naïve patients, at least 18 years of age and presenting with NVAF will be considered eligible for participation in this study only after the decision to treat with rivaroxaban has been made by the treating physician.
  Interventions: Drug: Rivaroxaban (Xarelto,Bay 59-7939)

INTERVENTIONS:
Drug: Rivaroxaban (Xarelto,Bay 59-7939) — 15 mg and 20 mg (OD)

SUMMARY:
This study is planned to collect prospective data and evaluate the safety and effectiveness of rivaroxaban for the prevention of stroke and systemic embolism in Indian patients with NVAF when used in clinical practice under real-life conditions.

The study will be conducted in routine clinical practice settings. Approximately 1000 patients from India will be enrolled in this study. Patients will be observed for maximum period of 12 months after the start of Xarelto treatment or until it is no longer possible (e.g. lost to follow-up, death, withdrawal) before the end of the observation period.

The decision by the investigator to start with of Xarelto must be independent of the inclusion of a patient to the study.

ELIGIBILITY:
Inclusion Criteria:

* Patient should be an adult female or male, ≥18 years of age;
* Patient should be diagnosed with NVAF and initiated with rivaroxaban treatment for prevention of stroke or systemic embolism per investigator's routine treatment practice;
* Patient should not have received rivaroxaban in the past;
* Patient/patient's legally acceptable representative should be willing to provide written informed consent.

Exclusion Criteria:

* Patient has contraindications to receive rivaroxaban therapy according to local prescribing information;
* Patient is receiving anticoagulant therapy for indication other than NVAF and that needs to be continued as per discretion of treating physician;
* Patient is participating in an investigational program with interventions outside of routine clinical practice.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Female and male patients ≥18 years of age with a diagnosis of NVAF will be enrolled only after the decision for treatment with rivaroxaban has been made by the investigator.
Sampling Method: Non-Probability Sample
Enrollment: 504 (Actual)
Dates: Start 2019-10-03 (Actual); Primary Completion 2023-12-23 (Actual); Study Completion 2024-12-16 (Actual)

PRIMARY OUTCOMES:
Incidence of major bleeding events | Up to 18 months
  Major bleeding events include:
  * Fatal bleeding
  * Symptomatic bleeding in a critical area or organ
  * Bleeding causing a fall in hemoglobin level of 20 g/L (1.24 mmol/L) or more, or leading to transfusion of two or more units of whole blood or red cells.
    * Hemoglobin level; or
    * Need for transfusion of packed red blood cells or whole blood.
Incidence of treatment-emergent AEs | Up to 18 months
Incidence of treatment-emergent SAEs | Up to 18 months
Incidence of all-cause death | Up to 18 months
  Deaths will be adjudicated as either vascular (e.g., due to stroke, embolism, myocardial infarction, or arrhythmia) or non-vascular (e.g., malignancy or infection).

SECONDARY OUTCOMES:
Incidence of symptomatic thromboembolic events | Up to 18 months
  The date of thromboembolic events, manner in which thromboembolic events were managed in the routine practice setting, and their outcomes will be recorded.
  The thromboembolic events include:
  * Stroke and transient ischemic attack (TIA)
  * Systemic embolism
  * Myocardial infarction
Non-major bleeding events | Up to 18 months
  The date of non-major bleeding events, treatment approaches employed during non-major bleeding events, and the associated outcomes will be collected.
AE rates in the different NVAF risk factor categories | Up to 18 months
  Rates of AEs across patients with different baseline risk profiles for stroke or bleeding calculated using Congestive heart failure, Hypertension, Age, Diabetes mellitus, Stroke(CHADS2), Vascular disease, Age, Sex category (CHA2DS2-VASc), or Hypertension, Abnormal liver/renal function, Stroke history, Bleeding predisposition, Labile international normalized ratios, Elderly, Drug/alcohol usage (HAS-BLED).
SAE rates in the different NVAF risk factor categories | Up to 18 months
  Rates of SAEs across patients with different baseline risk profiles for stroke or bleeding calculated using Congestive heart failure, Hypertension, Age, Diabetes mellitus, Stroke (CHADS2), Vascular disease, Age, Sex category (CHA2DS2-VASc), or Hypertension, Abnormal liver/renal function, Stroke history, Bleeding predisposition, Labile international normalized ratios, Elderly, Drug/alcohol usage (HAS-BLED).
Treatment persistence with rivaroxaban | Up to 18 months
  Treatment persistence with rivaroxaban therapy will be defined as the absence of a gap of >60 days between two doses of rivaroxaban, without any switch to alternative anticoagulant. Reasons for any switch from or interruption of rivaroxaban therapy during the observation period will be collected and summarized.

CONTACTS AND LOCATIONS:
Locations (1):
- Sunshine Hospital, Secunderabad, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.